CLINICAL TRIAL: NCT01264042
Title: Iron Supplementation During Pregnancy and Non-Transferrin-Bound Iron (NTBI)
Acronym: NTBI_pw
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof., Swiss Federal Institute of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NTBI_pw
Record Dates: First submitted 2010-12-20; First posted 2010-12-21 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Pregnancy
Keywords: Iron Supplementation,; week 24 to 28 at study day
MeSH Terms: interventions — ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FeSo4 (Experimental)
  Interventions: Dietary Supplement: Ferrous Sulfate

INTERVENTIONS:
Dietary Supplement: Ferrous Sulfate — 60 mg with 200 mL water, single administration
  Other Names: FeSO4, Dr. Paul Lohmann, Emmerthal, Germany

SUMMARY:
Although the essential role of iron during pregnancy is well established, concerns have been raised that current iron supplements given routinely during pregnancy may also have harmful consequences, such as increased oxidative stress and enhanced risks of infection, pre-eclampsia and impaired glucose regulation. A potential mechanism for the production of adverse effects is the appearance of non-transferrin-bound iron after oral administration of iron supplements. Non-transferrin-bound iron is more readily available to pathogens and could promote injurious free radical reactions that might add to the oxidative stress of pregnancy.

The present study will determine if oral administration of 60 mg of iron as ferrous sulfate during the second trimester of pregnancy is followed by the appearance of non-transferrin-bound iron two hours later. The investigators will examine the influence of a variety of factors, including iron status and previous use of iron supplements. Detection of non-transferrin-bound iron after administration of an iron supplement to pregnant women would be an important new observation that could lead to re-evaluation of current methods of iron supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman
* Age 18 to 45 years
* singleton pregnancy
* between 24 and 28 of gestation (at study day)
* regular visits at prenatal clinic
* capability and willingness to comply with study protocol
* voluntary signed informed consent

Exclusion Criteria:

* Multiple pregnancy
* Acute or chronic disease or disorder
* Incapability of following the study protocol
* Homelessness
* Active drug/alcohol dependence or abuse history
* Currently participating in another clinical trial or having participated in another clinical trial during the last 3 months prior to the beginning of this study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
NTBI | Change between baseline and 2 hours
  The primary variables are NTBI values determined at baseline and two hours after the intake of 60 mg ferrous sulfate, which will allow to determine the effect of the iron supplement on NTBI formation.

SECONDARY OUTCOMES:
Iron Status and History of Iron Supplements | baseline
  The secondary variables are iron status (Hb, ferritin, transferrin receptor) and the history of use of iron supplements. The results of NTBI measurements will be analyzed in relation to iron status and use of iron supplements.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Krafft, Dr., Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland